CLINICAL TRIAL: NCT04609566
Title: A Phase 2 Study of Brentuximab Vedotin in Combination With Pembrolizumab in Participants With Metastatic Solid Malignancies
Brief Title: Brentuximab Vedotin With Pembrolizumab in Metastatic Solid Tumors
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seagen, a wholly owned subsidiary of Pfizer (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Organization: Seagen Inc. (Industry)
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGN35-033; C5691005 (Other: Alias Study Number)
Record Dates: First submitted 2020-10-23; First posted 2020-10-30 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Melanoma; Non-small Cell Lung Cancer; Squamous Cell Carcinoma of the Head and Neck
Keywords: Seattle Genetics
MeSH Terms: conditions — Melanoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck | interventions — Brentuximab Vedotin; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Combination Therapy (Experimental): brentuximab vedotin + pembrolizumab
  Interventions: Drug: brentuximab vedotin; Drug: pembrolizumab

INTERVENTIONS:
Drug: brentuximab vedotin — 1.8 mg/kg given into the vein (IV; intravenously) every 3 weeks
  Other Names: ADCETRIS
Drug: pembrolizumab — 200 mg given intravenously every 3 weeks
  Other Names: KEYTRUDA®

SUMMARY:
This trial will find out whether brentuximab vedotin and pembrolizumab work together to treat different types of cancer. There will be several different types of cancer studied in the trial. The cancer must have spread to other parts of the body (metastatic).

The study will also find out what side effects occur. A side effect is anything the treatment does besides treat cancer.

This is a multi-cohort study.

ELIGIBILITY:
Inclusion Criteria

* Participants must have

  * Metastatic squamous or nonsquamous non-small cell lung cancer (NSCLC) (without known targetable EGFR, ALK, ROS1, or BRAF mutations) who either

    * a) have not yet received frontline therapy for metastatic disease and without prior exposure to anti PD-1/PD-L1 or
    * b) are relapsed/refractory with progression on anti PD-1/PD therapy.
  * Relapsed/refractory metastatic cutaneous melanoma (regardless of mutation status) with progression on a PD-1 inhibitor
  * Metastatic head and neck squamous cell carcinoma (HNSCC) who have not yet received frontline therapy for metastatic disease and without prior exposure to a PD-1/PD-L1 inhibitor.
* Cohorts 1-4 only: Melanoma participants must be currently on PD-1 checkpoint inhibitor (CPI) therapy (e.g. nivolumab or pembrolizumab) or had their last dose of PD-1 CPI containing therapy as the last previous line of therapy within 90 days prior to enrollment; PD-1 CPI therapy must be the immediate prior line of treatment.
* Cohorts 1-4 only: Participants must have progressed on treatment with an anti-PD-1 monoclonal antibody (mAb) administered either as monotherapy, or in combination with other CPIs or other therapies. PD-1 treatment progression is defined by meeting all of the following criteria.

  * Have received at least 2 doses of an approved PD-1 inhibitor.
  * Have demonstrated disease progression (PD) after a PD-1 inhibitor as defined by RECIST v1.1.

    * Progressive disease has been documented within 90 days from the last dose of PD-1 inhibitor.
    * Participants with melanoma will need iRECIST confirmation of progression with a second assessment at least four weeks after the initial date of progressive disease
    * NSCLC participants on PD-1 inhibitor containing therapy for less than 90 days will need iRECIST confirmation of progression at least 4 weeks after the initial date of progressive disease
* Tumor tissue sample obtained within 3 months prior to enrollment is required, and no systemic anticancer therapy given after the sample was obtained.
* An Eastern Cooperative Oncology Group (ECOG) Performance Status score of equal or less than 1

Exclusion Criteria

* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Prior immunosuppressive chemotherapy, any immunotherapy other than a PD-1 inhibitor within 4 weeks of first study drug dose.
* History of another malignancy within 3 years before the first dose of study drug or any evidence of residual disease from a previously diagnosed malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Confirmed objective response rate (ORR) based on investigator assessment using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) criteria | Up to approximately 2 years
  Confirmed ORR per RECIST v1.1 is defined as the proportion of participants whose best overall response is a confirmed complete response (CR) or partial response (PR) per RECIST v1.1.

SECONDARY OUTCOMES:
Duration of response (DOR) based on investigator assessment using RECIST v1.1 criteria | Up to approximately 3 years
  DOR per RECIST v1.1 is defined as the time from start of the first documentation of confirmed objective tumor response (CR or PR) per RECIST v1.1 to the first documentation of PD (per RECIST v1.1) or to death due to any cause, whichever comes first.
Progression-free survival (PFS) based on investigator assessment using RECIST v1.1 criteria | Up to approximately 3 years
  PFS is defined as the time from start of study treatment to first documentation of objective tumor progression (PD per RECIST v1.1), or to death due to any cause, whichever comes first.
ORR per iRECIST by investigator assessment | Up to approximately 2 years
  ORR per iRECIST is defined as the proportion of participants with confirmed CR or PR based on iRECIST guidelines
iDOR per iRECIST by investigator assessment | Up to approximately 3 years
  DOR per iRECIST is defined as the time from first documentation of confirmed objective response (CR or PR) based on iRECIST guidelines by investigator assessment to the first documentation of confirmed objective tumor progression per iRECIST by investigator assessment, or to death due to any cause, whichever comes first.
iPFS per iRECIST by investigator assessment | Up to approximately 3 years
  iPFS is defined as the time from start of study treatment to the first documentation of confirmed objective tumor progression per iRECIST by investigator assessment, treatment discontinuation following the unconfirmed progression or death due to any cause, whichever comes first.
Incidence of adverse events (AEs) | Up to approximately 2 years
  National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. Analyses of AEs will be summarized with descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (81):
- United States (81):
  - Arizona Oncology Associates, PC - HOPE, Tucson, Arizona
  - Highlands Oncology Group, PA, Fayetteville, Arkansas
  - Highlands Oncology Group, PA, Rogers, Arkansas
  - Highlands Oncology Group, PA, Springdale, Arkansas
  - California Cancer Associates for Research and Excellence, Inc (cCARE), Encinitas, California
  - California Cancer Associates for Research and Excellence, Inc. cCARE, Fresno, California
  - The Angeles Clinic And Research Institute, A Cedars-Sinai Affiliate, Los Angeles, California
  - Cedars-Sinai Medical Center, Samuel Oschin Comprehensive Cancer Institute (SOCCI), Los Angeles, California
  - California Cancer Associates for Research and Excellence Inc (cCARE), San Marcos, California
  - The Angeles Clinic and Research Institute, A Cedars-Sinai Affiliate (Emergency Back-Up Only), Santa Monica, California
  - Rocky Mountain Cancer Centers, LLP, Aurora, Colorado
  - Clinical and Translational Research Center (CTRC), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Inpatient Pavilion (AIP), Aurora, Colorado
  - University of Colorado Hospital - Anschutz Outpatient Pavilion (AOP), Aurora, Colorado
  - University of Colorado Hospital-Anschutz Cancer Pavilion (ACP), Aurora, Colorado
  - Rocky Mountain Cancer Centers, LLP, Boulder, Colorado
  - Rocky Mountain Cancer Centers, LLP, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, LLP, Denver, Colorado
  - Rocky Mountain Cancer Centers, LLP, Lakewood, Colorado
  - Rocky Mountain Cancer Centers, LLP, Littleton, Colorado
  - Rocky Mountain Cancer Centers, LLP, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, LLP, Longmont, Colorado
  - Rocky Mountain Cancer Centers, LLP, Pueblo, Colorado
  - Rocky Mountain Cancer Centers, LLP, Thornton, Colorado
  - Northwestern Medical Group, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - The University of Kansas Cancer Center, Investigational Drug Services, Westwood, Kansas
  - The University of Kansas Cancer Center, Westwood, Kansas
  - Norton Cancer Institute Downtown, Louisville, Kentucky
  - Norton Hospital, Louisville, Kentucky
  - Norton Audubon Hospital, Louisville, Kentucky
  - Norton Cancer Institute, Audubon Hospital Campus, Louisville, Kentucky
  - Norton Brownsboro Hospital, Louisville, Kentucky
  - Norton Cancer Institute, Brownsboro Hospital Campus, Louisville, Kentucky
  - Minnesota Oncology Hematology PA, Burnsville, Minnesota
  - Minnesota Oncology Hematology PA, Coon Rapids, Minnesota
  - Minnesota Oncology Hematology PA, Edina, Minnesota
  - Minnesota Oncology Hematology PA, Fridley, Minnesota
  - Minnesota Oncology Hematology PA, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA, Maplewood, Minnesota
  - Minnesota Oncology Hematology PA, Minneapolis, Minnesota
  - Minnesota Oncology Hematology PA, Plymouth, Minnesota
  - Minnesota Oncology Hematology PA, Saint Paul, Minnesota
  - Minnesota Oncology Hematology PA, Woodbury, Minnesota
  - Nebraska Medicine - Bellevue Medical Center, Bellevue, Nebraska
  - Nebraska Medicine, Omaha, Nebraska
  - Nebraska Medicine - Village Pointe, Omaha, Nebraska
  - University Of Nebraska Medical Center, Omaha, Nebraska
  - New York Oncology Hematology, P.C., Albany, New York
  - New York Oncology Hematology, P.C., Clifton Park, New York
  - Oncology_Hematology Care Clinical Trials,LLC, Cincinnati, Ohio
  - Oncology_Hematology Care Clinical Trials,LLC, Fairfield, Ohio
  - Toledo Clinic Cancer Center, Toledo, Ohio
  - Oncology Associates of Oregon, P.C., Eugene, Oregon
  - Texas Oncology - Central South, Austin, Texas
  - Texas Oncology - Central South (Balcones Dr), Austin, Texas
  - Texas Oncology - Central South (James Casey), Austin, Texas
  - Texas Oncology-DFW, Dallas, Texas
  - Texas Oncology - Fort Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology-DFW, Fort Worth, Texas
  - Oncology Consultants, PA, Houston, Texas
  - US Oncology Investigational Product Center (IPC), Irving, Texas
  - US Oncology Investigational Products Center (IPC), Irving, Texas
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Blacksburg, Virginia
  - Inova Schar Cancer Institue Infusion Pharmacy, Fairfax, Virginia
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Oncology & Hematology Associates of Southwest Virginia Inc., Low Moor, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - VCU Health Stony Point, Richmond, Virginia
  - Massey Cancer Center Clinical & Translational Research Lab, Richmond, Virginia
  - Tissue and Data Acquisition and Analysis Core (TDAAC), Richmond, Virginia
  - VCU Health- Adult Outpatient Pavilion (AOP) Investigational Drug Services, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Roanoke, Virginia
  - Oncology and Hematology Associates of Southwest Virginia, Inc., DBA Blue Ridge Cancer Care, Salem, Virginia
  - VCU Health Community Memorial Hospital, South Hill, Virginia
  - VCU Health Tappahannock Hospital, Tappahannock, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, INC., Wytheville, Virginia
  - Fred Hutchinson Cancer Care Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=SGN35-033